CLINICAL TRIAL: NCT00278512
Title: High Dose Immune Suppression With Hematopoietic Stem Cell Support in Refractory Vasculitis, Necrotizing Vasculitis, Neurovascular Behcet's Disease, and Sjogren's Syndrome
Brief Title: Hematopoietic Stem Cell Support in Vasculitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No participant enrolled over five years. No plan to continue the study.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAD Vasculitis.Auto2002
Record Dates: First submitted 2006-01-15; First posted 2006-01-18 (Estimated); Results first posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2017-06

CONDITIONS: Vasculitis
MeSH Terms: conditions — Vasculitis | interventions — Cyclophosphamide; thymoglobulin; Granulocyte Colony-Stimulating Factor; Filgrastim; Alemtuzumab; fludarabine; fludarabine phosphate; Tacrolimus; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous Stem Cell Transplant (Experimental): Autologous Stem Cell Transplant will be performed on eligible patients
  Interventions: Biological: Autologous Stem Cell Transplant; Biological: Allogeneic Stem Cell Transplant; Drug: Cyclophosphamide; Drug: ATG (rabbit); Drug: G-CSF; Drug: Mesna
- Allogeneic Stem Cell Transplant (Experimental): Allogeneic Stem Cell Transplant will be performed on eligible patients
  Interventions: Biological: Allogeneic Stem Cell Transplant; Drug: Cyclophosphamide; Drug: G-CSF; Drug: Campath-1h; Drug: Fludarabine; Drug: Tacrolimus; Drug: Mesna

INTERVENTIONS:
Biological: Autologous Stem Cell Transplant — Autologous Hematopoietic Stem Cell Transplant will be performed after conditioning
  Other Names: AutologousHematopoietic Stem Cell Transplantation
  Arms: Autologous Stem Cell Transplant
Biological: Allogeneic Stem Cell Transplant — Allogeneic Stem Cell Transplant will be performed after conditioning
  Other Names: Allogeneic Hematopoietic Stem Cell Transplantation
Drug: Cyclophosphamide — Causes prevention of the cell division
  Other Names: Cytoxan, Neosar
Drug: ATG (rabbit) — A rabbit polyclonal antibody to lymphocyte
  Other Names: Thymoglobulin
  Arms: Autologous Stem Cell Transplant
Drug: G-CSF — Hematopoietic growth factor
  Other Names: Neupogen
Drug: Campath-1h — Humanized monoclonal antibody against CD52 antigen
  Other Names: Alemtuzumab
  Arms: Allogeneic Stem Cell Transplant
Drug: Fludarabine — inhibits DNA synthesis or repair
  Other Names: Fludara
  Arms: Allogeneic Stem Cell Transplant
Drug: Tacrolimus — immune suppressive drug
  Other Names: FK506, PROGRAF
  Arms: Allogeneic Stem Cell Transplant
Drug: Mesna — Mesna is a drug used to protect the bladder from the effects of the chemotherapy drugs
  Other Names: Mesnex

SUMMARY:
The systemic vasculitis is a wide-ranging group of diseases that are characterized by the presence of blood vessel inflammation (1). Despite this common feature, each type of vasculitis has a unique variety of clinical manifestations that influences its degree of disease severity and ultimately its management. Immunosuppressive therapy forms the foundation of treatment for almost all forms of systemic vasculitis.

The systemic necrotizing vasculitis (SNV) are a subset of vasculitis with significant morbidity and mortality (2). The SNV are Wegener's granulomatosis, allergic angiitis and granulomatosis (AAG) (also known as Churg-Strauss syndrome), polyarteritis nodosum (PAN), microscopic polyangiitis (MPA), and overlap syndrome. In spite of modern therapeutic immune suppressive agents, there remains a not inconsequential morbidity and mortality associated with SNV. The current standard therapy for SNV is chronic oral cyclophosphamide (1-3 mg/kg/day) and corticosteroids (3-6). Transplant doses of cyclophosphamide at 200 mg/kg infused over 4 days is the most common worldwide transplant regimen for systemic lupus erythematosus (SLE) (7). Like SLE, SNV are cyclophosphamide responsive disease. We, therefore, propose a trial of high dose cyclophosphamide with anti-thymocyte globulin (ATG) for patients with SNV.

DETAILED DESCRIPTION:
Selection of High Dose Immunosuppressive Therapy and Autologous HSCT Strategy for this Trial

Selection of the Regimen for High-Dose Immunosuppressive Therapy Cyclophosphamide with ATG (Cy/ATG) is a common conditioning regimen with two decades of experience in the treatment of aplastic anemia and has been used safely without reported mortality in the treatment of autoimmune diseases such as systemic lupus erythematosus and rheumatoid arthritis. Cy/ATG not only has less acute toxicity, it has less chronic side effects. Cy/ATG is not associated with late malignancies or cataracts. Cyclophosphamide and anti-thymocyte globulin (horse or rabbit ATG) and rituximab are potent immunosuppressive agents. Rituximab and ATG contribute additional immunosuppression without additional cytotoxicity. Rituximab and ATG given shortly pre-transplant will contribute to the elimination of host T lymphocytes that survive cyclophosphamide or that contaminate the CD34+selected graft. SLE, an autoimmune disease responsive to cyclophosphamide, responds well to a Cy/ATG/rituximab conditioning regimen. For these reasons, Cy/ATG/rituximab will be the conditioning regimen utilized in this study.

To justify any new therapy such as HSCT, the risk of dying from the disease must be higher than that expected from its treatment, or the morbidities associated with the disease must justify the treatment risks. Autologous stem cell transplantation has a mortality of 1-3% in breast cancer patients using intense conditioning regimens with multiple alkylating agents, and up to 10-15% in patients with lymphomas and other malignancies. The latter patients usually have been heavily treated before transplant and the accumulation of treatment toxicities is thought to play a role in their increased transplant-related mortality. Cyclophosphamide and ATG/rituximab have been used to transplant of extremely ill patients with systemic lupus erythematosus and multiple organ dysfunction at Northwestern University without mortality.

Since patients in this study are earlier in the disease course, a conditioning regimen that has historically been associated with less toxicity will be employed. The regimen will be Cyclophosphamide at 200 mg/kg with ATG 5.5 mg/kg and rituximab 1000 mg divided over 2 doses. Cyclophosphamide 200mg/kg with or without ATG has been used safely and effectively in a variety of autoimmune diseases including systemic lupus erythematosus, rheumatoid arthritis, and aplastic anemia. Rabbit ATG will be used instead of equine ATG due to the lower incidence of hypersensitivity and fever with rabbit ATG compared to equine.

Method of Harvesting Stem Cells Based on the experience of the pilot studies, the current protocol will mobilize stem cells with cyclophosphamide and granulocyte-colony stimulating factor (G-CSF), and collect stem cells by apheresis, with subsequent bone marrow harvest performed only if needed to supplement the peripheral blood stem cells (PBSC). Based on experience of autoimmune flares in patients receiving G-CSF alone for mobilization (56), patients will be mobilized with cyclophosphamide 2.0 g/m2 and G-CSF 10 mcg /kg.

Regimen for Autologous HSCT

Cyclophosphamide Cyclophosphamide is an active agent in patients with a wide variety of malignancies. It is used frequently in the therapy of lymphoid malignancies and has potent immunosuppressive activity. It is frequently used as a cytotoxic and immunosuppressive agent in patients undergoing marrow transplants and as a treatment for patients with autoimmune diseases. It is an alkylating agent that requires hepatic metabolism to the active metabolites, phosphoramide mustard and acrolein. These active metabolites react with nucleophilic groups. It is available as an oral or intravenous preparation. Bioavailability is 90% when given orally. The half-life of the parent compound is 5.3 hours in adults, and the half-life of the major metabolite phosphoramide mustard is 8.5 hours. Liver or renal dysfunction will lead to prolonged serum half-life. CY is administered intravenously at a dosage of 50 mg/kg on each of two successive days (use adjusted ideal body weight if patient's actual body weight is greater than 100% ideal body weight). The major dose limiting side effect at high doses is cardiac necrosis. Hemorrhagic cystitis can occur and is mediated by the acrolein metabolite. This can be prevented by co-administration of MESNA or bladder irrigation. Other notable side effects include nausea, vomiting, alopecia, myelosuppression and SIADH. Refer to institutional manuals for more information about administration, toxicity and complications.

Rabbit-Derived Anti-Thymocyte Globulin (ATG) Rabbit-derived anti-thymocyte globulin (ATG) is a gamma globulin preparation obtained from hyperimmune serum of rabbits immunized with human thymocytes. ATG has been used predominately in solid organ transplant immunosuppressive regimens. ATG is a predominantly lymphocyte-specific immunosuppressive agent. It contains antibodies specific to the antigens commonly found on the surface of T cells. After binding to these surface molecules, ATG promotes the depletion of T cells from the circulation through mechanisms, which include opsonization and complement-assisted, antibody- dependent, cell-mediated cytotoxicity. The plasma half-life ranges from 1.5-12 days. ATG is administered intravenously at a dose of 0.5 mg/kg recipient body weight on day -6 and a dose of 1.0 mg/kg recipient body weight on days -5, -4, -3, -2 and -1. Unlike equine ATG, rabbit ATG does not require a pre-infusion skin test to check for hypersensitivity. Methylprednisolone 1 gram will be given before every dose of ATG. Additional medications such as diphenhydramine may be given at the discretion of the attending physician. Although rare, the major toxicity is anaphylaxis. Chills, fever, pruritus or serum sickness may occur.

Regimen for allogeneic HSCT

Cyclophosphamide (Cytoxan) Cyclophosphamide (CY) is administered intravenously at a dosage of 50 mg/kg on each of four successive days (use adjusted ideal body weight if patient's actual body weight is greater than 100% ideal body weight). The major dose limiting side effect at high doses is cardiac necrosis. Hemorrhagic cystitis can occur and is mediated by the acrolein metabolite. This can be prevented by co-administration of MESNA or bladder irrigation. Other notable side effects include nausea, vomiting, alopecia, myelosuppression and SIADH. Refer to institutional manuals for more information about administration, toxicity and complications.

Fludarabine Fludarabine phosphate is rapidly dephosphorylated to 2-fluoro-ara-A and then phosphorylated intracellularly by deoxycytidine kinase to the active triphosphate, 2-fluoro-ara-ATP. This metabolite appears to act by inhibiting DNA polymerase alpha, ribonucleotide reductase and DNA primase, thus inhibiting DNA synthesis. The mechanism of action of this antimetabolite is not completely characterized and may be multi-faceted.

Phase I studies in humans have demonstrated that fludarabine phosphate is rapidly converted to the active metabolite, 2-fluoro-ara-A, within minutes after intravenous infusion. Consequently, clinical pharmacology studies have focused on 2-fluoro-ara-A pharmacokinetics. After the five daily doses of 25 mg 2-fluoro-ara-AMP/m2 to cancer patients infused over 30 minutes, 2-fluoro-ara-A concentrations show a moderate accumulation. During a 5-day treatment schedule, 2-fluoro-ara-A plasma trough levels increased by a factor of about 2. The terminal half-life of 2-fluoro-ara-A was estimated as approximately 20 hours. In vitro, plasma protein binding of fludarabine ranged between 19% and 29%.

CAMPATH Campath-1H is a humanized fusion protein that is directed to CD52 antigen that is expressed on all lymphocytes, monocytes and macrophages. It has very potent immunosuppressive property and is effective for prevention of graft-versus-host disease. 30 mg/day of CAMPATH will be given intravenously over 2 hours on days -4, -3 and -2. The most commonly reported adverse reactions are infusion reactions fever, chills, hypotension, urticaria, nausea, rash, tachycardia, dyspnea), cytopenias (neutropenia, lymphopenia, thrombocytopenia, anemia), and infections (CMV viremia, CMV infection, other infections). In clinical trials, the frequency of infusion reactions was highest in the first week of treatment. Other commonly reported adverse reactions include vomiting, abdominal pain, insomnia and anxiety. The most commonly reported serious adverse reactions are cytopenias, infusion reactions, and immunosuppression/infections. About 30 minutes before the patient gets Campath, he/she will be given other medications (such as acetaminophen or diphenhydramine, given orally, not IV) to help reduce side effects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 16 to 60 years old at the time of pretransplant evaluation.
* 2. An established diagnosis of systemic necrotizing vasculitis (Wegener's granulomatous, polyarteritis nodosum (PAN), allergic angiitis granulomatous (AAG, also known as Churg Strauss syndrome), microscopic polyangiitis (MPA), or overlap syndrome)Temporal arteritis, or mixed cryoglobulinemia or primary central nervous system vasculitis AND failure of corticosteroids and any of the following at least 6 months of oral or IV cytoxan, rituximab, or cellcept. (Failure defined as: a) patients with a high disease activity and involvement of internal organs as measured by increased FFS > 2 and/or BVAS > 20, or b) patients who develop recurrent flares with subsequent progressive organ damage.)

OR

Neurovascular Behcets with recurrent oral and/or genital lesions confirmed by culture to be herpes negative, MRI findings consistent with CNS vasculitis, recurrent neurological symptoms, and clinical confirmation by a Neurologist (e.g., Dr. Rama Gourimeni) AND failure of at least 3 months of oral or IV cytoxan.

OR

Pulmonary or neurovascular Sjogrens with positive SSA/SSB confirmed by a rheumatologist and neurologist (if CNS involved) or pulmonologist (if lungs involved) and either recurrent neurologic attacks or progressive pulmonary compromise (dyspnea on exertion, decreased DLCO or CT findings of active disease) despite at least 6 months of intravenous monthly pulse cyclophosphamide.

* 3. Patient eligibility must be confirmed by two Rheumatologists. For patients with neurovascular Behcets, eligibility need only be confirmed by a neurologist.
* 4. A minimum CD34+ cell dose of 2.0 x 10e6/kg post-selection.

Exclusion Criteria:

* 1. Significant end organ damage such as:

  1. LVEF <40% or deterioration of LVEF during exercise test on MUGA or echocardiogram unless due to active disease.
  2. Untreated life-threatening arrhythmia.
  3. Active ischemic heart disease or heart failure.
  4. DLCO < 40% of predicted value unless due to active disease.
  5. Serum creatinine > 2.5 mg/dl, unless due to active disease.
  6. Liver cirrhosis, transaminases >3x of normal limits, or bilirubin >2.0 unless due to Gilberts disease.
* 2. HIV positive.
* 3. Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment.
* 4. Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer will be considered on an individual basis.
* 5. Positive pregnancy test, inability or unable to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
* 6. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
* 7. Inability to give informed consent.
* 8. Active infection, excluding asymptomatic bacteruria or vaginal candidiasis.
* 9. Active hepatitis B (HBSAg positive) or active hepatitis C (PCR positive blood lymphocytes).

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2003-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Autologous Stem Cell Transplant | Allogeneic Stem Cell Transplant
Started | 7 | 0
Completed | 6 | 0
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous Stem Cell Transplant | Allogeneic Stem Cell Transplant | Total
Number analyzed (Participants) | 7 | 0 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 0 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.43 (12.03) |  | 40.43 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 |  | 7

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Survival
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous Stem Cell Transplant | Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 7 | 0
Participants | 6 | 0

ADVERSE EVENTS:
Time Frame: 6 months, 1 year, then yearly for at least 5 years post transplant
Arm/Group | Autologous Stem Cell Transplant | Allogeneic Stem Cell Transplant
All-Cause Mortality (participants affected / at risk) | 1/7 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/0
Other Adverse Events (participants affected / at risk) | 2/7 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Stem Cell Transplant (N=7) | Allogeneic Stem Cell Transplant (N=0)
CMV Hepatitis (Infections and infestations) | 1 (1) | 0 (0) — One participant died of CMV hepatitis.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Stem Cell Transplant (N=7) | Allogeneic Stem Cell Transplant (N=0)
Swine flu (Infections and infestations) | 1 (1) | 0 (0) — One patient diagnosed with swine flu, requiring transient face mask oxygen and recovered.
Aspergillus (Infections and infestations) | 1 (1) | 0 (0) — One patient 4 years after transplant relapsed and was started on actemra. After 2 years of actemra ( a TNF inhibitor) patient developed aspergillus
Pseudomonas pneumonia (Infections and infestations) | 1 (1) | 0 (0) — One patient 4 years after transplant relapsed and was started on actemra. After 2 years of actemra ( a TNF inhibitor) patient developed pseudomonas pneumonia.
bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) — Two years after transplant had bowel obstruction due to pre transplant surgical scars-
Pulmonary Embolus (Cardiac disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small numbers of subjects enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes